CLINICAL TRIAL: NCT02985749
Title: A Pilot Study of Oxytocin for the Treatment of Social Impairment in Individuals With High Functioning Autism Spectrum Disorder
Brief Title: A Study of Oxytocin for the Treatment of Social Impairment in Individuals With High Functioning Autism Spectrum Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Gagan Joshi, Medical Director, Bressler Program for Autism Spectrum Disorders, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016P002148
Record Dates: First submitted 2016-11-17; First posted 2016-12-07 (Estimated); Results first posted 2023-08-16 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Autism Spectrum Disorder; Pervasive Developmental Disorder; ASD; PDD
Keywords: Autism Spectrum Disorders; Pervasive Developmental Disorder; ASD; PDD; Oxytocin; Syntocinon; Social Impairment; Treatment
MeSH Terms: conditions — Autism Spectrum Disorder; Child Development Disorders, Pervasive | interventions — Oxytocin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oxytocin- Participants ages 12-17 (Experimental): Intranasal Oxytocin (brand name Syntocinon) will be administered daily (for a total daily dose of 48 IU) for 8 weeks.
  Interventions: Drug: Intranasal Oxytocin
- Oxytocin- Participants ages 18-55 (Experimental): Intranasal Oxytocin (brand name Syntocinon) will be administered daily (for a total daily dose of 48 IU) for 8 weeks.
  Interventions: Drug: Intranasal Oxytocin

INTERVENTIONS:
Drug: Intranasal Oxytocin — This study is examining the short-term efficacy and tolerability of intranasal oxytocin for the treatment of social impairment in youths and adults with high-functioning ASD (HF-ASD).
  Other Names: Syntocinon

SUMMARY:
This study is an 8-week pilot trial with oxytocin nasal spray (Syntocinon) as a treatment for social impairment in children and adults with high functioning autism spectrum disorders (ASD). The investigators hypothesize that oxytocin will be safe, tolerable, and effective in improving social deficits in individuals with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 12 and 55 years of age.
* Meets the DSM-5 diagnostic criteria for Autism Spectrum Disorder (ASD) as established by clinical diagnostic interview
* At least moderate severity of ASD impairment as measured by a raw score of ≥85 on the SRS
* Participants and their parent/guardian must be able to speak and understand English sufficiently to comprehend the nature of the study and to allow for the completion of all study procedures required per protocol.
* Subjects and their parent/guardian must be considered reliable reporters. They must understand the nature of the study and must sign an IRB-approved informed consent form before initiation of any study procedures. Subjects and their parent/guardian must have a level of understanding sufficient to communicate with the investigator and study coordinator, and to cooperate with all tests and examinations required by the protocol.
* Each subject and their parent/guardian must understand the nature of the study and provide written informed assent/consent.
* Subjects with mood, anxiety, or disruptive behavior disorders will be allowed to participate in the study provided they do not meet any exclusionary criteria.
* If the subject is sexually active, he/she must agree to use an acceptable form of birth control during the study. These include:
* Abstinence (no sexual contact)
* A barrier method (diaphragm plus spermicide or a condom plus spermicide) in addition to one of the following methods:
* Consistent use of an approved birth control pill
* Birth control patch
* Injected contraceptives
* Intrauterine device (IUD)

Exclusion Criteria:

* Impaired intellectual functioning and/or impaired spoken language.
* Clinically unstable psychiatric conditions or any serious medical illness, which will be assessed by study clinicians during the psychiatric interview and medical history review. If the clinical assessment suggests a psychiatric or medical condition demanding acute clinical attention, then the subject will be excluded from participating in the trial.
* Clinically unstable psychiatric conditions.
* Any serious medical illness
* Pregnant or nursing females.
* Known hypersensitivity to oxytocin.
* Severe allergies or multiple adverse drug reactions.
* A non-responder or history of intolerance to oxytocin, after treatment at adequate doses as determined by the clinician.
* Subjects with significant nasal pathology (including atrophic rhinitis, recurrent nose bleeds, and history of hypophysectomy).
* Clinically abnormal baseline laboratory values falling significantly outside of the standard reference ranges for a basic metabolic screen.
* Investigator and his/her immediate family defined as the investigator's spouse, parent, child, grandparent, or grandchild.
* Currently enrolled or recently participated (within the past 6 months) in a clinical trial of intranasal oxytocin.

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gagan Joshi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Cambridge, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxytocin- Participants Ages 12-17: Participants ages 12-17 enrolled to receive oxytocin treatment
  Intranasal Oxytocin (brand name Syntocinon) will be administered daily (for a total daily dose of 48 IU) for 8 weeks.
  Intranasal Oxytocin: This study is examining the short-term efficacy and tolerability of intranasal oxytocin for the treatment of social impairment in youths and adults with high-functioning ASD (HF-ASD).
- Oxytocin- Participants Ages 18-55: Participants ages 18-55 enrolled to receive oxytocin treatment
  Intranasal Oxytocin (brand name Syntocinon) will be administered daily (for a total daily dose of 48 IU) for 8 weeks.
  Intranasal Oxytocin: This study is examining the short-term efficacy and tolerability of intranasal oxytocin for the treatment of social impairment in youths and adults with high-functioning ASD (HF-ASD).
Period: Overall Study
Arm/Group | Oxytocin- Participants Ages 12-17 | Oxytocin- Participants Ages 18-55
Started | 2 | 5
Completed | 2 | 3
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin- Participants Ages 12-17 | Oxytocin- Participants Ages 18-55 | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 0 | 2
  Between 18 and 65 years | 0 | 5 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.5 (2.1) | 30.0 (8.7) | 25.3 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 5 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in ASD Symptoms Social Responsiveness Scale 2 (SRS-2) Scale From Baseline to Week 8
Description: Change in ASD symptoms as measured by change from baseline on the Social Responsiveness Scale 2 (SRS-2) scale.
  The SRS-2 is a 65-item rating scale completed that is used to measure the severity of autism spectrum symptoms as they occur in natural settings. The SRS-2 School Age form is completed by a parent or guardian for patients ages 9-17 and the SRS-2 Adult Self-report is completed by patients ages 18-59. Total raw scores range from 0 to 195, with higher scores indicating increased symptom severity.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Oxytocin- Participants Ages 12-17 | Oxytocin- Participants Ages 18-55
Number analyzed (Participants) | 2 | 3
scores on a scale | -39.5 (12) | -29 (9.8)

ADVERSE EVENTS:
Time Frame: 8 weeks (from baseline to end of study)
Arm/Group | Oxytocin- Participants Ages 12-17 | Oxytocin- Participants Ages 18-55
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 1/2 | 3/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxytocin- Participants Ages 12-17 (N=2) | Oxytocin- Participants Ages 18-55 (N=5)
Ear infection (Ear and labyrinth disorders) | 0 (0) | 1 (3)
Foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Faint/dizzy after blood drawn (Nervous system disorders) | 0 (0) | 1 (1)
Drowsiness (Nervous system disorders) | 0 | 1 (1)
Allergy (Immune system disorders) | 1 (1) | 0 (0)
Increased sex drive (Psychiatric disorders) | 0 (0) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT02985749/Prot_SAP_000.pdf